CLINICAL TRIAL: NCT00067470
Title: Study of Recombinant Human N-acetylgalactosamine 4-sulfatase (rhASB) in Patients With MPS VI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASB-03-05
Record Dates: First submitted 2003-08-20; First posted 2003-08-25 (Estimated); Results first posted 2009-08-17 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-12

CONDITIONS: Mucopolysaccharidosis VI
MeSH Terms: conditions — Mucopolysaccharidosis VI | interventions — N-Acetylgalactosamine-4-Sulfatase

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- rhASB (Active Comparator)
  Interventions: Drug: N-acetylgalactosamine 4-sulfatase

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: N-acetylgalactosamine 4-sulfatase
  Other Names: rhASB
  Arms: rhASB

SUMMARY:
The purpose of the study is to evaluate the ability of rhASB versus placebo to enhance endurance in patients with Mucopolysaccharidosis VI (MPS VI), as evidenced by an increase in the number of meters walked in the 12 minute walk test at Week 24 compared with baseline.

ELIGIBILITY:
Inclusion Criteria

* Patient consent
* Patient must be seven years of age or older
* Patient must have documented biochemical or genetic proof of MPS VI
* The patient must be able to walk independently at least 5 meters and no more than 270 meters in the first 6 minutes, or no more then 400 meters total in 12 minutes, in the screening 12-minute walk test
* If female of childbearing potential, patient must have a negative pregnancy test

Exclusion Criteria

* Patient is under consideration for or has undergone a successful bone marrow transplant (BMT)
* Patient refuses or is unable to complete all screening evaluations
* Pregnant or lactating patient
* Patient has received an investigational drug within 30 days prior to study enrollment
* Patient has been previously treated with rhASB
* Patient has a medical condition, serious intercurrent illness, or other extenuating circumstance that may significantly confound study results or decrease study compliance
* The patient has clinically significant spinal cord compression
* The patient has known hypersensitivity to rhASB or to components of the active or placebo test solutions

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2003-09; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Locations (1):
- BioMarin Pharmaceutical Inc., Novato, California, United States

REFERENCES:
- [Derived] Tandon PK, Kakkis ED. The multi-domain responder index: a novel analysis tool to capture a broader assessment of clinical benefit in heterogeneous complex rare diseases. Orphanet J Rare Dis. 2021 Apr 19;16(1):183. doi: 10.1186/s13023-021-01805-5. PMID 33874971
- See also: Related Info — http://www.bmrn.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Locations:Oakland, CA, USA Mainz, Germany Manchester, England Porto Alegre, Brazil Lyon, France Porto, Portugal
  Study Duration: 24 weeks
  First enrollment: 21 July 2003
  Last Dose Given: 1 April 2004
  Last Assessment: 8 April 2004
Groups:
- rhASB: Intravenous (IV) recombinant human arylsulfatase(rhASB) at 1.0 mg/kg
- Placebo: Intravenous (IV) placebo solution at a volume equivalent to that needed for a 1.0 mg/kg dose of rhASB
Period: Overall Study
Arm/Group | rhASB | Placebo
Started | 19 | 20
Completed | 19 | 19
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rhASB | Placebo | Total
Number analyzed (Participants) | 19 | 20 | 39
Age Continuous [Mean (Standard Deviation); unit: years] | 13.7 (6.47) | 10.7 (4.35) | 12.2 (5.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 7 | 6 | 13
Race/Ethnicity, Customized [Number; unit: participants]
  White, non-Hispanic | 15 | 9 | 24
  Hispanic | 1 | 3 | 4
  Black | 1 | 2 | 3
  Asian | 1 | 1 | 2
  Indigenous | 1 | 1 | 2
  Other | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 2 | 4 | 6
  Germany | 4 | 4 | 8
  United Kingdom | 3 | 3 | 6
  Brazil | 4 | 4 | 8
  France | 2 | 3 | 5
  Portugal | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 12-minute Walk Test at 24 Weeks
Description: Number of meters walked in 12 minutes at week 24 minus number of meters walked in 12 minutes at baseline
Time Frame: baseline and 24 weeks
Population: The efficacy analysis included all subjects except one from the placebo group who withdrew from the study prior to the week 24 assessment.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | rhASB | Placebo
Number analyzed (Participants) | 19 | 19
meters | 109 (154) | 26 (122)
Statistical Analysis 1: Comparison: rhASB vs Placebo; Test type: Superiority or Other; p = 0.025, Regression, Linear; Mean Difference (Net) = 92, 95% CI [11 to 172], Standard Error of Mean 40

2. Secondary Outcome: Change From Baseline in 3-minute Stair Climb at 24 Weeks
Description: Number of stairs climbed per minute in 3 minutes at 24 weeks minus number of stairs climbed per minute in 3 minutes at baseline
Time Frame: baseline and 24 weeks
Population: The efficacy analysis included all subjects except one from the placbo group who withdrew from the study prior to the week 24 assessment.
Measure: Mean (Standard Deviation); unit: stairs/min
Arm/Group | rhASB | Placebo
Number analyzed (Participants) | 19 | 19
stairs/min | 7.4 (9.9) | 2.7 (6.9)
Statistical Analysis 1: Comparison: rhASB vs Placebo; Test type: Superiority or Other; p = 0.053, Regression, Linear; The raw data were adjusted for the observed differences in baseline between the groups and fitted to a longitudinal repeated measures linear model; Mean Difference (Net) = 5.7, 95% CI [-0.1 to 11.5], Standard Error of Mean 2.9

3. Secondary Outcome: Change From Baseline in Urinary GAG (uGAG) at 24 Weeks
Description: Glycosaminoglycan (GAG) level measured in urine
Time Frame: baseline and 24 weeks
Population: Baseline uGAG level was measured for 19 rhASB-treated subjects and 20 placebo-treated subjects. However, uGAG levels at 24 weeks were measured for 19 rhASB-treated subjects and 19 placebo-treated subjects, because 1 placebo-treated subject withdrew from the study before week 24.
Measure: Mean (Standard Deviation); unit: micrograms per mg creatinine
Arm/Group | rhASB | Placebo
Number analyzed (Participants) | 19 | 19
micrograms per mg creatinine
  Baseline Urinary GAG Level | 346 (128) | 330 (114)
  24-week Urinary GAG Level | 85 (35) | 317 (80)

ADVERSE EVENTS:
Arm/Group | rhASB | Placebo
Serious Adverse Events (participants affected / at risk) | 3/19 | 4/20
Other Adverse Events (participants affected / at risk) | 19/19 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhASB (N=19) | Placebo (N=20)
Abdominal Strangulated Hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Apnoea (Infections and infestations) | 1 (1) | 0 (0)
Cardiac failure congestive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Convulsion (Infections and infestations) | 1 (1) | 1 (1)
Corneal lesion (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ileus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (1)
Obstructive airways disorder (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Viral infection (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhASB (N=19) | Placebo (N=20)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 6 (6)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abscess oral (Infections and infestations) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Acute tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Anasarca (General disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Application site erythema (General disorders) | 1 (1) | 0 (0)
Areflexia (Nervous system disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 7 (7)
Asthenia (General disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Bladder pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Blister (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood phosphorus increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Bloody discharge (General disorders) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 2 (2)
Cardiomegaly (Cardiac disorders) | 0 (0) | 1 (1)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Cervical myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 3 (3) | 1 (1)
Clonus (Nervous system disorders) | 1 (1) | 0 (0)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 4 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Corneal opacity (Eye disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6)
Dental caries (Infections and infestations) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 6 (6)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 2 (2) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 8 (8) | 4 (4)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Exanthem (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 1 (1) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1)
Face oedema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 1 (1) | 2 (2)
Gait abnormal (General disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 1 (1)
Granuloma (General disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 8 (8) | 12 (12)
Hearing impaired (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 3 (3)
Hepatosplenomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hernia pain (General disorders) | 2 (2) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hip deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 2 (2)
Hydrocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hyperaemia (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 3 (3) | 3 (3)
Infusion site pain (General disorders) | 1 (1) | 2 (2)
Intestinal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Keratoconjunctivitis sicca (Eye disorders) | 0 (0) | 2 (2)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Malaise (General disorders) | 2 (2) | 0 (0)
Mass (General disorders) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 5 (5)
Nausea (Gastrointestinal disorders) | 4 (4) | 5 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Oral Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 5 (5) | 4 (4)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Pain (General disorders) | 5 (5) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (8)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Paresis (Nervous system disorders) | 1 (1) | 2 (2)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (1)
Petechiae (Vascular disorders) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (3) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 4 (4)
Poor venous access (Vascular disorders) | 1 (1) | 3 (3)
Post procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 8 (8) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Rigors (General disorders) | 4 (4) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 4 (4)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Nervous system disorders) | 1 (1) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Sputum abnormal (Investigations) | 1 (1) | 0 (0)
Suprapubic pain (General disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thirst (General disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tic (Psychiatric disorders) | 0 (0) | 1 (1)
Tongue oedema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Tooth Disorder (Gastrointestinal disorders) | 0 (0) | 2 (2)
Tooth discoloration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 7 (7)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vaginitis (Infections and infestations) | 0 (0) | 1 (1)
Ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (6) | 7 (7)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication of the results shall be made by Sponsor in a joint publication. If such a multi-center publication is not submitted within 12 months after conclusion of the study, the PI may publish the results from their site individually, subject however to comply with the other terms of the agreement.